CLINICAL TRIAL: NCT03270501
Title: Efficacy of Golimumab in Early Axial Spondyloarthritis in Relation to Gut Inflammation, an Early Remission Induction Study
Brief Title: Efficacy of Golimumab in Early Axial Spondyloarthritis in Relation to Gut Inflammation
Acronym: GO-GUT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); the Flanders Institute for Biotechnology (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO-GUT trial
Record Dates: First submitted 2017-08-18; First posted 2017-09-01 (Actual); Results first posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-07

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Arm 1: Golimumab (Experimental)
  Interventions: Drug: Golimumab

INTERVENTIONS:
Drug: Golimumab — Axial spondyloarthritis patients who don't have a good treatment response on 2 NSAIDs, will be treated with golimumab. After remission, the therapy will be stopped.
  All patients will undergo a ileocoloscopy at baseline and, if positive, at time of remission.
  Other Names: ileocoloscopy

SUMMARY:
The hypothesis of the study is that the presence of (subclinical) gut inflammation at baseline in patients with early active axial spondyloarthritis predisposes to a more severe disease defined as more need to use anti-tumor necrosis factor α therapy and a shorter time to relapse after stopping anti-tumor necrosis factor α therapy after obtaining sustained clinical remission. Overall, the investigators hypothesize that subclinical gut inflammation is an important predictor in therapy response and outcome. These data could provide better insights into the complex interactions between gut and joint inflammation and guide the physicians in the therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a diagnosis of axSpA and classified according to ASAS criteria.
* Subject has at least 3 months and maximum 1 year (almost) daily chronic back pain.
* Subject has an active disease defined as a positive MRI (according to ASAS definition) or elevated CRP (in patients who are HLA-B27+) and an ASDAS score > 2.1 (at least high disease activity).

Exclusion Criteria:

* Full anti-inflammatory dose of NSAIDs for more than 4 weeks for the duration of the axSpA symptoms.
* Prior exposure to any biologic therapy with a potential therapeutic impact on SpA, including anti-TNF therapy.
* Exposure to disease-modifying drugs (DMARDSs; i.e. methotrexate and sulfasalazine) in the last 3 months before the ileocolonoscopy.
* Exposure to systemic corticosteroid treatment in the last 14 days before the ileocolonoscopy.
* Infection(s) requiring treatment with intravenous antibiotics/antivirals/antifungals within 30 days prior to the baseline visit or oral antibiotics/antivirals/antifungals within 14 days prior to the baseline visit.
* Have a known hypersensitivity to human immunoglobulin proteins or other components of golimumab.
* History of central nervous system (CNS) demyelinating disease or neurologic symptoms suggestive of CNS demyelinating disease.
* History of listeriosis, histoplasmosis, chronic of active hepatitis B infection, hepatitis C infection, human immunodeficiency virus (HIV) infection, immunodeficiency syndrome, chronic recurring infections or active tuberculosis.
* Have a history of, or concurrent, chronic heart failure, including medically controlled, asymptomatic congestive heart failure.
* Evidence of dysplasia or history of malignancy (including lymphoma and leukemia) other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma or localized carcinoma in situ of the cervix.
* Have received, or are expected to receive, any live virus or bacterial vaccination within 3 months prior to the first administration of study agent, during the trial, or within 6 months after the last administration of study agent.
* Positive pregnancy test at screening.
* Female subjects who are breast-feeding or considering becoming pregnant during the study.
* Female subjects who do not use contraceptives.
* History of clinically significant drug or alcohol abuse in the last 12 months.
* Clinically significant abnormal screening laboratory results as evaluated by the investigator.
* Positive rheumatoid factor (RF) or anti-cyclic citrullinated peptide (anti-CCP) antibody at screening if the titers are crossing 3 times the upper limit of the normal.
* Subject with diagnosis and current symptoms of fibromyalgia.
* Any medical or psychological condition that, in the opinion of the investigator, could jeopardize or compromise the subject's ability to participate in this study.

Ages: 18 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Elewaut, Principal Investigator — University Ghent
Locations (3):
- Belgium (3):
  - Imelda Bonheiden, Bonheiden, Antwerpen
  - Ghent University Hospital, Ghent, B - Belgium
  - Reuma Instituut Hasselt, Hasselt, Limburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dougados M, Baeten D. Spondyloarthritis. Lancet. 2011 Jun 18;377(9783):2127-37. doi: 10.1016/S0140-6736(11)60071-8. PMID 21684383
- [Background] Mielants H, Veys EM, Cuvelier C, De Vos M, Botelberghe L. HLA-B27 related arthritis and bowel inflammation. Part 2. Ileocolonoscopy and bowel histology in patients with HLA-B27 related arthritis. J Rheumatol. 1985 Apr;12(2):294-8. PMID 3875721
- [Background] Van Praet L, Van den Bosch FE, Jacques P, Carron P, Jans L, Colman R, Glorieus E, Peeters H, Mielants H, De Vos M, Cuvelier C, Elewaut D. Microscopic gut inflammation in axial spondyloarthritis: a multiparametric predictive model. Ann Rheum Dis. 2013 Mar;72(3):414-7. doi: 10.1136/annrheumdis-2012-202135. Epub 2012 Nov 8. PMID 23139267

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: November 2017 - December 2022 across 3 centres:
  * Gent University Hospital
  * Imelda Hospital in Bonheiden
  * Jessa Hospital in Hasselt
Groups:
- Arm 1: NSAIDs With Possible Step-up to Golimumab: NSAIDs: All patients fulfilling the inclusion criteria will be treated according to the current recommendations for the management of axial spondyloarthritis, i.e. with 2 courses of NSAIDs. If sufficient response is acheived, the patients will continue receiving NSAIDs and after sustained remission, the therapy will be stopped. If therapy with NSAIDs provides insufficient control of disease activity, switch to therapy with Golimumab will be made.
  Golimumab: Patients who did not have a good treatment response to 2 NSAIDs, will be treated with golimumab sc 50mg/4 weeks. After sustained remission, the therapy will be stopped.
  All patients will undergo a ileocoloscopy at baseline and, if positive, at time of remission.
Period: Overall Study
Arm/Group | Arm 1: NSAIDs With Possible Step-up to Golimumab
Started | 64
Treatment Protocol Initiated | 58
Completed | 55
Not Completed | 9
Not completed — Screen failure | 6
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Patients included in the trial and for whom the treatment protocol was initiated.
Arm/Group | Arm 1: NSAIDs With Possible Step-up to Golimumab
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 2
Ankylosing Spondylitis Disease Activity Score (ASDAS)-CRP [Mean (Standard Deviation); unit: units on a scale] — ASDAS is a composite index to assess disease activity in axSpA. ASDAS parameters: 1) Total back pain 2) Patient global 3) Peripheral pain/swelling 4) Duration of morning stiffness 5) CRP in mg/L: ASDAS calculation: 0.121 × total back pain + 0.110 × patient global + 0.073 × peripheral pain/swelling + 0.058 × duration of morning stiffness + 0.579 × Ln(max(CRP,2)+1). Parameters 1-4 are reported by patients on a visual analogue score ranging from 0 to 10. Data from five variables combine to yield a score (minimum 0.636 to no defined upper limit), higher scores indicate higher disease activity.
  units on a scale | 3.0 (0.9)
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) [Mean (Standard Deviation); unit: units on a scale] — BASDAI is a measure of disease activity which was calculated based on 6 separate questionnaire items that were answered by the patients using visual analogue scale scales with range 0-10. A weighted average was performed, where items 5 and 6 had a weight of 0.5 whereas items 1, 2, 3 and 4 had a weight of 1. Range is from 0 to 10, with 10 indicating more severe disease activity.
  units on a scale | 4.5 (1.5)
Bath Ankylosing Spondylitis Functional index (BASFI) [Mean (Standard Deviation); unit: units on a scale] — BASFI is a measure of physical function which was calculated based on 10 separate questionnaire items that were answered by the patients using visual analogue scales with range 0-10, an average across 10 items was calculated. The range is 0-10 with 10 indicating that the level of physical functioning is more severely affected.
  units on a scale | 3.0 (2.2)
Positive for HLA-B27 (%) [Count of Participants; unit: Participants] | 50
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.3 (4.7)
Time from diagnosis [Median (Standard Deviation); unit: days] — Time from the first diagnosis of axial spondyloarthritis to enrollment in the trial
  days | 37 (18)
Assessment of SpondyloArthritis international Society (ASAS) criteria: Inflammatory Back Pain [Count of Participants; unit: Participants] — IBP according to experts: four out of five of the following parameters present: (1) age at onset less than 40 years, (2) insidious onset, (3) improvement with exercise, (4) no improvement with rest, (5) pain at night (with improvement upon getting up). (Reference: Ann Rheum Dis 2009;68:777-83)
  Participants | 51
Assessment of SpondyloArthritis international Society (ASAS) criteria: Arthritis [Count of Participants; unit: Participants] — Documented past or present active synovitis diagnosed by a doctor.
  Participants | 5
Assessment of SpondyloArthritis international Society (ASAS) criteria: Good response to NSAIDs [Count of Participants; unit: Participants] — Patient-reported effect of treatment with over-the-counter administered NSAIDs taken against axial spondyloarthritis symptoms.
  Participants | 44
Assessment of SpondyloArthritis international Society (ASAS) criteria: Heel enthesitis [Count of Participants; unit: Participants] — Heel enthesitis: past or present spontaneous pain or tenderness at examination at the site of the insertion of the Achilles tendon or plantar fascia at the calcaneus. (Reference: Ann Rheum Dis 2009;68:777-83)
  Participants | 3
Assessment of SpondyloArthritis international Society (ASAS) criteria: Psoriasis [Count of Participants; unit: Participants] — Documented past or present psoriatic skin or nail lesions diagnosed by a doctor.
  Participants | 0
Assessment of SpondyloArthritis international Society (ASAS) criteria: Uveitis [Count of Participants; unit: Participants] — Documented past or present anterior uveitis, diagnosed by an ophthalmologist. (Reference: Ann Rheum Dis 2009;68:777-83)
  Participants | 0
Assessment of SpondyloArthritis international Society (ASAS) criteria: Dactylitis [Count of Participants; unit: Participants] — Documented past or present dactylitis diagnosed by a doctor. (Reference: Ann Rheum Dis 2009;68:777-83)
  Participants | 0
Assessment of SpondyloArthritis international Society (ASAS) criteria: Inflammatory bowel disease [Count of Participants; unit: Participants] — Documented past or present inflammatory bowel disease diagnosed by a doctor. (Reference: Ann Rheum Dis 2009;68:777-83)
  Participants | 1
Assessment of SpondyloArthritis international Society criteria: Elevated C-reactive protein [Count of Participants; unit: Participants] — Measured within 3 months priort to study inclusoon or at baseline and temporally associated with patient's complaints emergence of CRP above upper normal limit in the presence of back pain, after exclusion of other causes for elevated CRP concentration. (Reference: Ann Rheum Dis 2009;68:777-83)
  Participants | 24
Assessment of SpondyloArthritis international Society criteria: Family history of spondyloarthritis [Count of Participants; unit: Participants] — Patient reported presence in first-degree or second-degree relatives of any of the following: (a) ankylosing spondylitis, (b) psoriasis, (c) uveitis, (d) reactive arthritis, (e) inflammatory bowel disease. (Reference: Ann Rheum Dis 2009;68:777-83)
  Participants | 22
CRP (mg/mL) [Mean (Standard Deviation); unit: mg/mL] | 7.6 (11)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Achieving Sustained Clinical Remission
Description: The proportion of patients who completed the trial and achieved Ankylosing Spondylitis Disease Activity Score (ASDAS-CRP) < 1.3 recorded on 2 consecutive visits with at least 12 weeks interval. ASDAS-CRP was measured at every study visit, i.e. baseline, week 2, week 4, week 16, week 28, week 40 and week 52. The study endpoint could earliest be achieved at visit week 28.
Time Frame: Upon end of trial for individual patient, between 28 and 52 weeks.
Population: Patients who completed the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: NSAIDs With Possible Step-up to Golimumab
Number analyzed (Participants) | 55
Participants | 34

2. Secondary Outcome: The Proportion of Patients With Healed Lesions of the Intestinal Mucosa
Description: According to the protocol, every patient underwent ileocolonoscopy at baseline to screen for macroscopic and microscopic (histopathologic analysis of endoscopic biopsies) signs of inflammation. If baseline ileocolonoscopy was protocolled as positive, the patient would undergo a second ileocolonoscopic assessment at the timepoint of reaching sustained clinical remission (study endpoint). The outcome measure is the proportion of patients with a negative second ileocolonoscopy.
Time Frame: At reaching primary outcome (between week 24 and week 52)
Population: At baseline ileocolonoscopy, macroscopic lesions justifying a repeated ileocolonoscopy at a later timepoint were found in only 1 patient. For this patient, pathologic findings present at baseline assessment were also found during the second assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: NSAIDs With Possible Step-up to Golimumab
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events data was collected between the first dose administration of trial medication and the last trial related activity (through study completion, between 24 weeks and 52 weeks). Medical events that occurred between signing of the Informed Consent and the first intake of trial medication were documented as medical and surgical history section and concomitant diseases.
Description: All adverse events and serious adverse events were recorded in the patient's file and in the Case Report Form. Adverse Events were defined as any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Arm/Group | Arm 1: NSAIDs With Possible Step-up to Golimumab
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 19/58
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: NSAIDs With Possible Step-up to Golimumab (N=58)
Nasopharyngitis (Infections and infestations) | 14 (16) — Viral or bacterial upper respiratory tract infection, including confirmed SARS-CoV-2 infections.
Gastroenteritis (Infections and infestations) | 4 (4) — Gastroenteritis
Otitis (Infections and infestations) | 3 (3) — External (otitis externa) or middle (otitis media) ear infection

LIMITATIONS AND CAVEATS:
The trial included 64 of initially anticipated 147 patients, which impacts downstream analyses which were powered for a larger group.

The baseline prevalence of gut inflammation in the studied patient population was lower than anticipated. Therefore primary objective of the study (to evaluate whether there is a higher need of anti-TNFα treatment in patients with gut inflammation compared to those without) could not be adressed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT03270501/Prot_SAP_000.pdf